CLINICAL TRIAL: NCT06003699
Title: Mindfulness Training in the Medical Health Care System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Amishi Jha, Professor, University of Miami
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 20230690
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Burnout, Professional; Stress; Emotion Regulation
MeSH Terms: conditions — Burnout, Professional; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness training group (Experimental): Participants will receive 4 weeks of mindfulness-based training and then continue to have access to the mindfulness training exercise throughout the second training interval.
  Interventions: Behavioral: Search Inside Yourself (SIY) program
- Wait-list Control Group (Active Comparator): Participants will not receive 4 weeks of mindfulness-based training during the first training interval; they will receive 4 weeks of mindfulness training during the second training interval.
  Interventions: Behavioral: Search Inside Yourself (SIY) program

INTERVENTIONS:
Behavioral: Search Inside Yourself (SIY) program — The present project involves the delivery of the Search Inside Yourself (SIY) program. The SIY Program is organized into 6 thematic modules. The first module introduces mindfulness and emotional intelligence and provides scientific evidence for the benefits of practicing mindfulness. The second module introduces Self-Awareness. The remaining four modules cover other domains based on Daniel Goleman's original framework of Emotional Intelligence: self-management, motivation, empathy, and leadership. Each module is associated with a set of practices, such as focused attention, body scan, journaling, empathic listening, and a Leadership Commitment exercise. The program will be delivered over 4 weeks, with one 3-hour session per week for a total of 12 hours that will take to complete all the modules.

SUMMARY:
The purpose of this study is to look at how mindfulness-informed emotional intelligence training may influence how participants think, feel, and act.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are between 18 and 80 years of age
2. Individuals who are fluent English speakers
3. Individuals who are able to adequately and independently use electronic devices, such as a laptop, computer, or tablet, and have Internet connection
4. Individuals who are willing and able to consent to participate in the study

Exclusion Criteria:

1. Individuals with an active and untreated mental health issue and/or hospitalization for psychological/mental health issues within the past month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Change in Positive Affect | Baseline, up to 11 weeks
  Positive Affect is assessed with the 5-item positive sub-scale from Positive and Negative Affect Schedule (PANAS). PANAS Positive has a range of scores from 5 to 25, with a higher score indicating a higher positive mood.
Change in Negative Affect | Baseline, up to 11 weeks
  Negative Affect is assessed with the 5-item positive sub-scale from Positive and Negative Affect Schedule (PANAS). PANAS Negative has a range of scores from 5 to 25, with a higher score indicating a higher negative mood.
Change in Perceived Stress | Baseline, up to 11 weeks
  Perceived stress is assessed with the 4-item Perceived Stress Scale (PSS-4). PSS-4 has a range of scores from 0 to 16, with a higher score indicating a higher level of perceived stress.
Change in Decentering | Baseline, up to 11 weeks
  Decentering is assessed via the 11-item decentering sub-scale of the experience questionnaire (EQ-D). The decentering score ranges from 1 to 55, with a higher score indicating a higher level of decentering.
Change in Mindfulness | Baseline, up to 11 weeks
  Mindfulness is assessed with the 15-item short version of the Five Factor Mindfulness Questionnaire (FFMQ). The scores range from 15 to 75 with higher scores indicating greater levels of mindfulness.
Change in Leadership Self-Awareness | Baseline, up to 11 weeks
  Leadership Self-Awareness is assessed with the 4-item self-awareness sub-scale from the Authentic Leadership Questionnaire (ALQ). Each item is rated on a 5-point Likert Scale ranging from 0 ("not at all") to 4 ("frequently"), and higher scores indicate greater self-awareness.
Change in Workplace Emotional Intelligence | Baseline, up to 11 weeks
  Workplace Emotional Intelligence is assessed with the 16-item Workplace Emotional Intelligence Profile Scale (WEIPS). Each item is rated on a scale from 1("strongly disagree") to 7 ("strongly"), and higher scores indicate greater emotional intelligence.

SECONDARY OUTCOMES:
Change in Attentional Performance | Baseline, up to 11 weeks
  The Sustained Attention Response Task (SART) is used to assess attentional performance and mind wandering (i.e., off-task thinking which is typically self-generated and compromises the performance of the task at hand). SART has a range of scores from 0 to 1 with a higher score indicating better accuracy when completing the task.
Change in Depression and Anxiety | Baseline, up to 11 weeks
  Depression and anxiety is assessed with the 4-item Patient Health Questionnaire (PHQ-4) Each item is rated from 0 ("not at all") to 3 ("nearly every day"), and ratings are summed together. PHQ-4 has a range of scores from 0 to 12, with higher scores indicating higher levels of depression and anxiety.
Change in Burnout | Baseline, up to 11 weeks
  Burnout will be assessed with the 12-item Burnout Assessment Tool (BAT-12). Each item is rated on a 5-point Likert scale from 0 ("never") to 5 ("always"). Ratings are then averaged on a scale of 0 to 5, where a higher score indicates greater burnout.
Change in Flourishing | Baseline, up to 11 weeks
  Flourishing will be assessed using the 8-item Flourishing Scale. Each item is rated on a 7-point Likert scale from 0 ("Strongly disagree") to 7 ("Strongly agree"). Ratings are then averaged with higher scores representing greater psychological resources and strengths.
Change in Sleep | Baseline, up to 11 weeks
  Sleep problems will be assessed with one question assessing the overall quality of the participants' sleep. The item is rated on a 4-point Likert scale. Scores range from 0 to 3 with a higher score indicating lower quality sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Amishi Jha, PhD, Principal Investigator — University of Miami
Locations (1):
- McLaren Health Care Corporation, Grand Blanc, Michigan, United States

IPD SHARING:
Plan to Share IPD: No